CLINICAL TRIAL: NCT02528071
Title: Prognostic Value of a Diaphragmatic Endurance Test in Patients With Amyotrophic Lateral Sclerosis : Impact and Prognosis. Single-center Prospective Pilot Study
Brief Title: Prognostic Value of a Diaphragmatic Endurance Test in Patients With Amyotrophic Lateral Sclerosis
Acronym: SLA
Status: Terminated | Type: Observational
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1308188; 2014-A00309-38 (Other: ANSM)
Record Dates: First submitted 2015-08-18; First posted 2015-08-19 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: ALS (Amyotrophic Lateral Sclerosis)
Keywords: Amyotrophic Lateral Sclerosis; ALS; Diaphragmatic Endurance Test
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: ALS patients performing measurements of maximal respiratory forces, diaphragmatic endurance during a diaphragmatic endurance test and phrenic nerve activity at the onset of the disease and repeated every 3 months up to respiratory failure or death
  Interventions: Other: Diaphragmatic endurance test
- Control: Healthy controls performing measurements of maximal respiratory forces, diaphragmatic endurance during a diaphragmatic endurance test and phrenic nerve activity. This arm will enable to establish reference values of IHT
  Interventions: Other: Diaphragmatic endurance test

INTERVENTIONS:
Other: Diaphragmatic endurance test — This consists of hyperventilation in a flask while maintaining the constant level of Carbon Dioxide (CO2). The patient will realize hyperventilation to increasing levels of Maximum Minute Ventilation (MMV), corresponding to increasing levels of respiratory rate, until exhaustion

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease which involves respiratory muscles and can lead at short term to respiratory failure. The occurrence of respiratory failure is associated with morbidity and an increased mortality. To date, respiratory muscle weakness is predicted from the reduction of vital capacity, maximal inspiratory force, nocturnal symptoms and hypercapnia. Even taken together, the predictive value of these indices is low.

The investigators hypothesize that an endurance test of diaphragmatic work would be more sensitive to respiratory muscle involvement than maximal respiratory force.

Consequently, the investigators assessed diaphragmatic performance through an isocapnic hyperventilation test (IHT) in patients at the onset of ALS and, then regularly up to the occurrence of respiratory failure. The investigators make the hypothesis that IHT will be altered earlier than maximal inspiratory force

ELIGIBILITY:
Inclusion Criteria for Patients :

* Older than 18 years old and younger than 80 years old
* ALS patient seen during the diagnostic assessment

Inclusion Criteria for control group :

* Older than 25 years old and younger than 80 years old
* No respiratory or neurologic active pathology

Exclusion Criteria for Patients :

* Bulbar ALS (inability to perform maximal respiratory maneuvers)
* Dementia
* Respiratory failure at diagnosis (arterial carbon dioxide partial pressure (pCO2) > 45 mmHg)
* Respiratory or neurologic active pathology

Exclusion Criteria for control group :

* Chest wall deformation with spirometric defect

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with ALS Healthly volonteers
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-09-29 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Endurance time | Day 1
  Difference in endurance time during the IHT between healthy controls and ALS patients when diagnosis is established

SECONDARY OUTCOMES:
Reference values of the diaphragmatic endurance test | Day 1
  Reference values of the diaphragmatic endurance test in healthy controls according to age, by 10 years range.
Reference values of phrenic nerve activity | Day 1
  Reference values of phrenic nerve activity in healthy controls according to age. It is measured with diaphragmatic Electromyogram by cervical electrical stimulation.
Slope of endurance time decrease | At Day 1 and every 3 months of follow-up (3 years)
  Slope of endurance time decrease with time in ALS patients measured during IHT
Amplitude of phrenic nerve | At Day 1 and every 3 months of follow-up (3 years)
  It is the relationship between phrenic nerve activity and diaphragmatic endurance in ALS patients
Latency of phrenic nerve | At Day 1 and every 3 months of follow-up (3 years)
  It is the relationship between phrenic nerve activity and diaphragmatic endurance in ALS patients

CONTACTS AND LOCATIONS:
Overall Officials: Frederic COSTES, MD PhD, Study Chair — CHU de Clermont-Ferrand; Isabelle COURT-FORTUNE, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No